CLINICAL TRIAL: NCT06096324
Title: Education and Employment Support for HIV Prevention in Young Adults (ENSPIRE)
Acronym: ENSPIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 23-1034; R01MD016815 (NIH)
Record Dates: First submitted 2023-10-09; First posted 2023-10-23 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-03

CONDITIONS: Economic Hardship; Condomless Sex; Utilization, Health Care
Keywords: HIV
MeSH Terms: conditions — Financial Stress; Unsafe Sex; Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Job announcements plus HIV prevention text messages, educational sessions, economic resources, and mentoring.
  Interventions: Behavioral: Job announcements plus HIV prevention text messages, educational sessions, economic resources, and mentoring.
- Control (Other): Job announcements only
  Interventions: Behavioral: Job announcements

INTERVENTIONS:
Behavioral: Job announcements plus HIV prevention text messages, educational sessions, economic resources, and mentoring. — Participants will receive job announcements plus HIV prevention text messages, educational sessions, economic resources, and mentoring.
  Arms: Intervention
Behavioral: Job announcements — Participants will receive job announcements only.
  Arms: Control

SUMMARY:
The study team will conduct a two-group study to examine the efficacy of implementing a combination intervention to improve economic stability and HIV preventive behaviors. The team will enroll approximately 500 young adults. Participants will be randomly assigned to one of two groups. The first group ("control") will receive text messages with information on job openings. The second group ("intervention") will receive text messages with information on job openings plus HIV prevention text messages, educational sessions on employment, income generation, and HIV prevention, economic resources, and mentoring.

DETAILED DESCRIPTION:
The study team will conduct a two-group study to examine the efficacy of implementing a combination intervention to improve economic stability and HIV preventive behaviors. The team will enroll approximately 500 young adults, aged 18 to 24, who are economically-vulnerable, sexually active, living in Baltimore, and have access to a mobile phone with text messaging. Participants will be recruited using respondent-driven sampling and be randomly assigned to one of two groups by cluster, equal to a seed and recruits. The first group ("control") will receive text messages with information on job openings. The second group ("intervention") will receive text messages with information on job openings plus HIV prevention text messages, educational sessions on employment, income generation, and HIV prevention, economic resources, and mentoring. Both groups will receive the assigned intervention for 12 weeks, equal to approximately 3 months. Data will be collected using participant surveys for one year at pre-intervention (Time 0), immediately post-intervention (Time 1, primary endpoint), and 6- and 12-months post-intervention (Time 2 to Time 3, longitudinal endpoints). Participants will undergo a baseline interview at the time of enrollment (Time 0) and be randomized to a group. Each group will receive the assigned activities for 12 weeks, at which point a follow-up interview will be conducted (Time 1, primary endpoint).

The study team will collect efficacy data pertaining to the following outcomes at T1 (Aim 1): (i) the mean economic stability score of participants in each group in the past six months (=primary outcome); (ii), the proportion of participants in each group who report one or more vaginal or anal sex acts without using a condom in the past six months (=secondary outcome); and (iii) the proportion of participants in each group who report PrEP continuum progressive movement of one or more stages in the past six months (=secondary outcome). All outcomes data will be collected using participant surveys.

The study team will also collect data on other pre-specified measures from T1 to T3 to characterize the primary and secondary aims (Aim 1), to assess differences in the efficacy of the intervention by sex and peer support (Aim 2), and to explore potential mediating factors over time (Aim 3). These other pre-specified measures include: (i) the proportion of participants in each group who report one or more paid hours of work in the past six months; (ii) the mean financial distress score of participants in each group in the past six months; (iii) the mean total money spent on HIV prevention activities of participants in each group in the past six months; (iv) the mean economic self-efficacy score of participants in each group in the past six months; (v) the proportion of participants in each group who report one or more other sexual risk behaviors associated with HIV acquisition in the past six months; (vi) the proportion of participants in each group who report one or more other care-seeking behaviors associated with HIV prevention in the past six months; (vii) the mean condom self-efficacy score of participants in each group in the past six months; (viii) the mean PrEP self-efficacy score of participants in each group in the past six months; (ix) the mean grit score of participants in each group in the past six months; and (x) the mean industriousness score of participants in each group in the past six months. All other pre-specified data will also be collected using participant surveys.

ELIGIBILITY:
Inclusion criteria are:

* Aged 18-24
* Economically-vulnerable in past 12 months
* Sexually active in past 12 months
* Living in Baltimore
* Has access to mobile phone with text messaging

Exclusion criteria are:

* Aged 17 or younger
* Older than 24 years
* Unwilling to provide consent for study participation

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Mean economic stability score of participants in each group in the past six months | Month 3
  The economic stability score of participants in each group in the past six months will be measured using a participant survey. The economic stability scale measures extent of economic stability and ranges from 0 to 64 with higher scores indicating a better outcome.

SECONDARY OUTCOMES:
Proportion of participants in each group who report one or more vaginal or anal sex acts without using a condom in the past six months | Month 3
  The proportion of participants in each group who report one or more vaginal or anal sex acts without using a condom in the past six months will be measured using a participant survey.
Proportion of participants in each group who report pre-exposure prophylaxis (PrEP) continuum progressive movement of one or more stages in the past six months | Month 3
  The proportion of participants in each group who report pre-exposure prophylaxis (PrEP) continuum progressive movement of one or more stages in the past six months will be measured using a participant survey. Participants will be assigned to one of nine stages based on their survey responses.

OTHER OUTCOMES:
Proportion of participants in each group who report one or more paid hours of work in the past six months | Month 3, Month 6, Month 12
  The proportion of participants in each group who report one or more paid hours of work in the past six months will be measured using a participant survey.
Mean financial distress score of participants in each group in the past six months | Month 3, Month 6, Month 12
  The mean financial distress score of participants in each group in the past six months will be measured using a participant survey. The financial distress scale measures extent of financial distress and ranges from 0 to 10 with higher scores indicating a worse outcome.
Mean total money spent on HIV prevention activities of participants in each group in the past six months | Month 3, Month 6, Month 12
  The mean total money spent on HIV prevention activities of participants in each group in the past six months will be measured using a participant survey.
Mean economic self-efficacy score of participants in each group in the past six months | Month 3, Month 6, Month 12
  The mean economic self-efficacy score of participants in each group in the past six months will be measured using a participant survey. The economic self-efficacy scale measures extent of economic self-efficacy and ranges from 0 to 16 with higher scores indicating a better outcome.
Proportion of participants in each group who report one or more other sexual risk behaviors associated with HIV acquisition in the past six months | Month 3, Month 6, Month 12
  The proportion of participants in each group who report one or more other sexual risk behaviors associated with HIV acquisition in the past six months will be measured using a participant survey.
Proportion of participants in each group who report one or more other care-seeking behaviors associated with HIV prevention in the past six months | Month 3, Month 6, Month 12
  The proportion of participants in each group who report one or more other care-seeking behaviors associated with HIV prevention in the past six months will be measured using a participant survey.
Mean condom self-efficacy score of participants in each group in the past six months | Month 3, Month 6, Month 12
  The mean condom self-efficacy score of participants in each group in the past six months will be measured using a participant survey. The condom self-efficacy scale measures extent of condom self-efficacy and ranges from 0 to 16 with higher scores indicating a better outcome.
Mean pre-exposure prophylaxis (PrEP) self-efficacy score of participants in each group in the past six months | Month 3, Month 6, Month 12
  The mean pre-exposure prophylaxis (PrEP) self-efficacy score of participants in each group in the past six months will be measured using a participant survey. The pre-exposure prophylaxis (PrEP) self-efficacy scale measures extent of PrEP self-efficacy and ranges from 0 to 14 with higher scores indicating a better outcome.
Mean grit score of participants in each group in the past six months | Month 3, Month 6, Month 12
  The mean grit score of participants in each group in the past six months will be measured using a participant survey. The grit scale measures extent of grit and ranges from 0 to 18 with higher scores indicating a better outcome.
Mean industriousness score of participants in each group in the last six months | Month 3, Month 6, Month 12
  The mean industriousness score of participants in each group in the last six months will be measured using a participant survey. The industriousness scale measures extent of industriousness and ranges from 0 to 26 with higher scores indicating a better outcome.
Mean economic stability score of participants in each group in the past six months | Month 6, Month 12
  The mean economic stability score of participants in each group in the past six months will be measured using a participant survey. The economic stability scale measures extent of economic stability and ranges from 0 to 64 with higher scores indicating a better outcome.
Proportion of participants in each group who report one or more vaginal or anal sex acts without using a condom in the past six months | Month 6, Month 12
  The proportion of participants in each group who report one or more vaginal or anal sex acts without using a condom in the past six months will be measured using a participant survey.
Proportion of participants in each group who report pre-exposure prophylaxis (PrEP) continuum progressive movement of one or more stages in the past six months | Month 6, Month 12
  The proportion of participants in each group who report pre-exposure prophylaxis (PrEP) continuum progressive movement of one or more stages in the past six months will be measured using a participant survey. Participants will be assigned to one of nine stages based on their survey responses.

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Jennings Mayo-Wilson, PhD MHS, Principal Investigator — University of North Carolina, Chapel Hill; Adriana Parker, MPH, Study Director — University of North Carolina, Chapel Hill
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data (IPD) will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: The IPD will be posted on a permanent online data repository within 36 months after study completion.
Access Criteria: There are no access criteria.